CLINICAL TRIAL: NCT04375007
Title: Correlation Between Self-efficacy, Fear of Movement, Empowerment, Enablement and Number of Visits to Physiotherapist for Patients With Musculoskeletal Disorders in Primary Health Care: A Feasibility Study
Brief Title: Factors Related to the Number of Visits to PT in PHC
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Number of visits to PT
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Physiotherapy; Musculoskeletal disorders; Self-efficacy; Empowerment; Enablement
MeSH Terms: conditions — Musculoskeletal Diseases; Empowerment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Routine care — Physiotherapy intervention in routine care

SUMMARY:
Musculoskeletal disorders can be a large burden on individuals, health care and social care systems. The aim was to assess the feasibility of performing a prospective study investigating whether self-efficacy, fear of movement, empowerment or enablement has any relation to the number of visits to physiotherapists among patients with a musculoskeletal disorder in primary health care. Design was apProspective study with consecutively selection including patients seeking physiotherapist for the first time for a musculoskeletal disorder. Primary outcome measure included operational and practical feasibility regarding recruitment of participants, use of questionnaires and key variables to be collected as part of the study.

DETAILED DESCRIPTION:
Background: Musculoskeletal disorders can be a large burden on individuals, health care and social care systems. Patients with musculoskeletal disorders are often treated by physiotherapists in primary health care. Psychosocial variables can be a significant obstacle to recover from musculoskeletal injuries.

The primary aim of this pilot study was to assess the feasibility of performing a prospective study investigating whether self-efficacy, fear of movement, empowerment or enablement has any relation to the number of visits to physiotherapist among patients with a musculoskeletal disorder in primary health care.

Methods: Prospective study with consecutively selection including patients seeking physiotherapist for the first time for a musculoskeletal disorder. Primary outcome measure included operational and practical feasibility regarding recruitment of participants, use of questionnaires and key variables to be collected as part of the study. Secondary outcomes included correlation between self-efficacy (Exercise Self-Efficacy Scale (ESES-S)), fear of movement (Tampa Scale for Kinesiophobia (TSK-SV)), empowerment (Making Decisions Scale ), enablement (Patient Enablement Instrument (PEI)) and number of visits to physiotherapist. Statistical analysis was done using IBM SPSS statistics version 24 with analysis of correlation using Spearman's rank correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who seek physiotherapist for the first time for a musculoskeletal disorder, are over 18 years of age and are able to read, write and understand Swedish.

Exclusion Criteria:

* Patients, who have visited physiotherapist previous for the same musculoskeletal disorder and/or are diagnosed with malignant diseases. Patients, who suffer from dementia, severe mental illness or other conditions making them not able to understand the information about the study and not able to fill in the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, visiting physiotherapist in primary health care in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | Through study completion, an average of 5 months
  Recruitment rate, time to recruit
Number of visits | Through study completion, an average of 5 months
  Count

SECONDARY OUTCOMES:
Exercise self-efficacy | At baseline
  Questionnarie
Kinesiophobia | At baseline
  Questionnarie
Empowerment | At baseline
  Questionnaire
Enablement | At baseline
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, PhD, Principal Investigator — Lund University
Locations (1):
- Primary Health Care Centre Åparken., Tyringe, Sweden

IPD SHARING:
Plan to Share IPD: No
This is not possible due to Swedish law